CLINICAL TRIAL: NCT00023699
Title: A Phase II Trial of ZD1839 (Iressa) (NSC# 715055) in the Treatment of Persistent or Recurrent Epithelial Ovarian or Primary Peritoneal Carcinoma
Brief Title: Gefitinib in Treating Patients With Recurrent or Persistent Ovarian Epithelial Cancer or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068852; GOG-0170C
Record Dates: First submitted 2001-09-13; First posted 2003-10-15 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2003-08

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Gefitinib

INTERVENTIONS:
Drug: gefitinib

SUMMARY:
RATIONALE: Biological therapies such as gefitinib may interfere with the growth of the tumor cells and may slow the growth of ovarian epithelial cancer or primary peritoneal cancer.

PURPOSE: Phase II trial to study the effectiveness of gefitinib in treating patients who have recurrent or persistent ovarian epithelial cancer or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor cytostatic activity of gefitinib, in terms of 6-month progression-free survival, in patients with persistent or recurrent ovarian epithelial or primary peritoneal carcinoma.
* Determine the nature and degree of toxicity in patients treated with this drug.
* Determine the partial and complete response rates in patients treated with this drug.
* Determine the duration of progression-free and overall survival in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral gefitinib once daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 22-60 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial or primary peritoneal carcinoma

  * Recurrent or persistent disease
* Must have had prior therapy with no more than 1 platinum-based chemotherapy regimen (e.g., carboplatin, cisplatin, or other organoplatinum compound) for primary disease
* Platinum-resistant or refractory

  * Treatment-free interval of less than 6 months after therapy with platinum-containing regimen OR
  * Progression during platinum-containing regimen OR
  * Platinum sensitive defined as treatment-free interval without disease progression for more than 6 months but less than 12 months after therapy with platinum-containing regimen
* At least 1 lesion measurable in at least 1 dimension

  * At least 20 mm by conventional techniques (e.g., palpation, plain x-ray, CT scan, or MRI) OR
  * At least 10 mm by spiral CT scan
* At least 1 target lesion outside a previously irradiated field
* Disease must be accessible to core needle biopsy
* Ineligible for higher priority GOG protocol

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* GOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No unstable cardiac disease
* No myocardial infarction within the past 6 months
* Coronary artery disease, congestive heart failure, and dysrhythmia allowed if on stable regimen for at least 3 months

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No sensory or motor neuropathy greater than grade 1
* No active corneal disease (e.g., keratoconjunctivitis)
* No active infection requiring antibiotics
* No evidence of bowel dysfunction that could be related to early bowel obstruction
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior immunological agents for the malignancy
* No concurrent anti-cancer immunotherapy

Chemotherapy:

* See Disease Characteristics
* No more than 1 additional prior cytotoxic chemotherapy regimen for recurrent or persistent disease
* No prior noncytotoxic chemotherapy for recurrent or persistent disease
* At least 3 weeks since prior chemotherapy for the malignancy and recovered
* No concurrent anti-cancer chemotherapy

Endocrine therapy:

* At least 1 week since prior anticancer hormonal therapy
* Concurrent hormone replacement therapy allowed
* No concurrent anti-cancer hormonal therapy

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy for the malignancy and recovered
* No prior radiotherapy to more than 25% of marrow-bearing areas
* No concurrent anti-cancer radiotherapy

Surgery:

* At least 4 weeks since prior surgery (except minor procedures under local anesthesia (e.g., central venous port placement)) and recovered

Other:

* At least 3 weeks since other prior therapy for the malignancy
* No prior gefitinib
* No other prior epidermal growth factor receptor inhibitors
* No prior anticancer therapy that would preclude study therapy
* No concurrent chlorpromazine
* No other concurrent investigational agents
* No other concurrent antineoplastic agents
* No concurrent CYP3A4-inducing agents, including phenytoin, carbamazepine, barbiturates, nafcillin, rifampicin, or St. John's Wort

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-08; Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell J. Schilder, MD, Study Chair — Fox Chase Cancer Center
Locations (53):
- United States (50):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Community Hospital of Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Medical Oncology Clinical Research Unit, Bethesda, Maryland
  - Tufts University School of Medicine, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Schneider Children's Hospital at North Shore, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Brookview Research, Inc., Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Fletcher Allen Health Care - Medical Center Campus, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- Australia New Zealand Gynaecological Oncology Trials Group, Camperdown, New South Wales, Australia
- Tom Baker Cancer Center - Calgary, Calgary, Alberta, Canada
- University of Birmingham, Birmingham, England, United Kingdom

REFERENCES:
- [Result] Schilder RJ, Sill MW, Chen X, Darcy KM, Decesare SL, Lewandowski G, Lee RB, Arciero CA, Wu H, Godwin AK. Phase II study of gefitinib in patients with relapsed or persistent ovarian or primary peritoneal carcinoma and evaluation of epidermal growth factor receptor mutations and immunohistochemical expression: a Gynecologic Oncology Group Study. Clin Cancer Res. 2005 Aug 1;11(15):5539-48. doi: 10.1158/1078-0432.CCR-05-0462. PMID 16061871